CLINICAL TRIAL: NCT05690230
Title: Improving the Patient Experience During Bone Marrow Biopsy/Aspiration (BMBA): Do Interventions Decrease Distress and Pain
Brief Title: Improving Patient Experience: BMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Daisy Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21G.1035; JT 18448 (Other: JeffTrial Number)
Record Dates: First submitted 2022-12-21; First posted 2023-01-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Bone Marrow Cancer; Leukemia; Lymphoma; Multiple Myeloma; Hematologic Cancer
MeSH Terms: conditions — Bone Marrow Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Two interventions will be trialed, each in parallel with a control group. The two phases will be done in sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1: Virtual reality (Experimental)
  Interventions: Other: Virtual reality
- Control 1 (No Intervention): Standard of care without change, in parallel with intervention 1: Virtual reality.
- Intervention 2: Environmental changes (Experimental)
  Interventions: Other: Environmental changes
- Control 2 (No Intervention): Standard of care without change, in parallel with intervention 2: Environmental changes.

INTERVENTIONS:
Other: Virtual reality — Patients will be provided with a wireless virtual reality headset that contains a guided meditation application. The application allows users to select their preferred music, visual setting, and a topic for meditation.
  Arms: Intervention 1: Virtual reality
Other: Environmental changes — A nature themed wall mural decal will be installed in the procedure room and the in-room computer will play music from Pandora. A selection of suggested stations will be provided, with the option for outside selections.
  Arms: Intervention 2: Environmental changes

SUMMARY:
This study seeks to determine if patients undergoing a bone marrow biopsy/aspiration (BMBA) procedure who receive distraction techniques have lower levels of distress and pain, and higher post-procedure satisfaction, compared to those receiving standard-of-care. Intervention 1 is guided meditation in a virtual reality (VR) headset. Intervention 2 is comprised of environmental changes to the room (via nature-themed decals) and music.

DETAILED DESCRIPTION:
This study seeks to determine if patients undergoing a bone marrow biopsy/aspiration (BMBA) procedure who receive distraction techniques have lower levels of distress and pain, and higher post-procedure satisfaction, compared to those receiving standard-of-care. Intervention 1 is guided meditation in a virtual reality (VR) headset. Intervention 2 is comprised of environmental changes to the room (via nature-themed decals) and music.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures
* Over 18 years of age
* Prior history of at least 1 (one) BMBA at Jefferson outpatient oncology office within the past 2 (two) years
* Visiting the Jefferson outpatient oncology office for a BMBA procedure during the study duration

Exclusion Criteria:

* Inability to read questions in English
* Inability to answer questions autonomously
* History of vertigo
* Legal blindness in both eyes
* Severe or profound hearing loss, or deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Distress score | Within 10 minutes pre-procedure
  The primary outcome will be reported on a scale of 0-10, based on the National Comprehensive Cancer Network (NCCN) Distress Thermometer, 0 signifying "no distress" and 10 signifying "extreme distress." This scale is standardly used with oncology patients to determine their distress levels-distress refers to "an unpleasant experience of a mental, physical, social, or spiritual nature. It can affect the way you think, feel, or act. Distress may make it harder to cope with having cancer, its symptoms, or its treatment."
Distress score | Within 10 minutes post-procedure
  The primary outcome will be reported on a scale of 0-10, based on the National Comprehensive Cancer Network (NCCN) Distress Thermometer, 0 signifying "no distress" and 10 signifying "extreme distress." This scale is standardly used with oncology patients to determine their distress levels-distress refers to "an unpleasant experience of a mental, physical, social, or spiritual nature. It can affect the way you think, feel, or act. Distress may make it harder to cope with having cancer, its symptoms, or its treatment."

SECONDARY OUTCOMES:
Pain intensity | Within 10 minutes pre-procedure
  To assess patient pain scores related to their BMBA procedure. This will be measured through the 0-10 Numeric Pain Intensity Scale, 0 signifying "no pain" and 10 signifying "the worst pain imaginable."
Pain intensity | Within 10 minutes post-procedure
  To assess patient pain scores related to their BMBA procedure. This will be measured through the 0-10 Numeric Pain Intensity Scale, 0 signifying "no pain" and 10 signifying "the worst pain imaginable."
Patient satisfaction | Within 10 minutes post-procedure
  To assess patient satisfaction with their procedure. This will be assessed through a patient satisfaction survey including Likert-type questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schweitzer M, Gilpin L, Frampton S. Healing spaces: elements of environmental design that make an impact on health. J Altern Complement Med. 2004;10 Suppl 1:S71-83. doi: 10.1089/1075553042245953. PMID 15630824
- [Background] Watts G, Khan A, Pheasant R. Influence of soundscape and interior design on anxiety and perceived tranquillity of patients in a healthcare setting. Applied Acoustics. 2016 Mar; 104:135-41.
- [Background] Ulrich RS. Effects of interior design on wellness: theory and recent scientific research. J Health Care Inter Des. 1991;3:97-109. PMID 10123973
- [Background] Laursen J, Danielsen A, Rosenberg J. Effects of environmental design on patient outcome: a systematic review. HERD. 2014 Summer;7(4):108-19. doi: 10.1177/193758671400700410. PMID 25303431
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899
- [Background] Iyendo TO, Uwajeh PC, Ikenna ES. The therapeutic impacts of environmental design interventions on wellness in clinical settings: A narrative review. Complement Ther Clin Pract. 2016 Aug;24:174-88. doi: 10.1016/j.ctcp.2016.06.008. Epub 2016 Jul 1. PMID 27502819
- [Background] Tsai HF, Chen YR, Chung MH, Liao YM, Chi MJ, Chang CC, Chou KR. Effectiveness of music intervention in ameliorating cancer patients' anxiety, depression, pain, and fatigue: a meta-analysis. Cancer Nurs. 2014 Nov-Dec;37(6):E35-50. doi: 10.1097/NCC.0000000000000116. PMID 24662723
- [Background] Danhauer SC, Vishnevsky T, Campbell CR, McCoy TP, Tooze JA, Kanipe KN, Arrington SA, Holland EK, Lynch MB, Hurd DD, Cruz J. Music for patients with hematological malignancies undergoing bone marrow biopsy: a randomized controlled study of anxiety, perceived pain, and patient satisfaction. J Soc Integr Oncol. 2010;8(4):140-147. PMID 24619452
- [Background] Thoma MV, Zemp M, Kreienbuhl L, Hofer D, Schmidlin PR, Attin T, Ehlert U, Nater UM. Effects of Music Listening on Pre-treatment Anxiety and Stress Levels in a Dental Hygiene Recall Population. Int J Behav Med. 2015 Aug;22(4):498-505. doi: 10.1007/s12529-014-9439-x. PMID 25200448
- [Background] Daniel E. Music used as anti-anxiety intervention for patients during outpatient procedures: A review of the literature. Complement Ther Clin Pract. 2016 Feb;22:21-3. doi: 10.1016/j.ctcp.2015.11.007. Epub 2015 Dec 1. PMID 26850800
- [Background] Speca M, Carlson LE, Goodey E, Angen M. A randomized, wait-list controlled clinical trial: the effect of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients. Psychosom Med. 2000 Sep-Oct;62(5):613-22. doi: 10.1097/00006842-200009000-00004. PMID 11020090
- [Background] Deng G, Cassileth BR. Integrative oncology: complementary therapies for pain, anxiety, and mood disturbance. CA Cancer J Clin. 2005 Mar-Apr;55(2):109-16. doi: 10.3322/canjclin.55.2.109. PMID 15761079
- [Background] Sander Wint S, Eshelman D, Steele J, Guzzetta CE. Effects of distraction using virtual reality glasses during lumbar punctures in adolescents with cancer. Oncol Nurs Forum. 2002 Jan-Feb;29(1):E8-E15. doi: 10.1188/02.ONF.E8-E15. PMID 11845217
- [Background] Espinoza M, Banos RM, Garcia-Palacios A, Cervera JM, Esquerdo G, Barrajon E, Botella C. Promotion of emotional wellbeing in oncology inpatients using VR. Stud Health Technol Inform. 2012;181:53-7. PMID 22954828
- [Background] Wiederhold BK, Gao K, Sulea C, Wiederhold MD. Virtual reality as a distraction technique in chronic pain patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):346-52. doi: 10.1089/cyber.2014.0207. PMID 24892196
- [Background] Bekelis K, Calnan D, Simmons N, MacKenzie TA, Kakoulides G. Effect of an Immersive Preoperative Virtual Reality Experience on Patient Reported Outcomes: A Randomized Controlled Trial. Ann Surg. 2017 Jun;265(6):1068-1073. doi: 10.1097/SLA.0000000000002094. PMID 27906757
- [Background] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Nanda U, Chanaud C, Nelson M, Zhu X, Bajema R, Jansen BH. Impact of visual art on patient behavior in the emergency department waiting room. J Emerg Med. 2012 Jul;43(1):172-81. doi: 10.1016/j.jemermed.2011.06.138. Epub 2012 Feb 9. PMID 22325555
- [Background] Harte R, Glynn L, Rodriguez-Molinero A, Baker PM, Scharf T, Quinlan LR, OLaighin G. A Human-Centered Design Methodology to Enhance the Usability, Human Factors, and User Experience of Connected Health Systems: A Three-Phase Methodology. JMIR Hum Factors. 2017 Mar 16;4(1):e8. doi: 10.2196/humanfactors.5443. PMID 28302594
- [Background] Devlin AS, Andrade CC, Carvalho D. Qualities of Inpatient Hospital Rooms: Patients' Perspectives. HERD. 2016 Apr;9(3):190-211. doi: 10.1177/1937586715607052. Epub 2015 Dec 14. PMID 26666814
- [Background] Satija A, Bhatnagar S. Complementary Therapies for Symptom Management in Cancer Patients. Indian J Palliat Care. 2017 Oct-Dec;23(4):468-479. doi: 10.4103/IJPC.IJPC_100_17. PMID 29123357
- [Background] Bani Mohammad E, Ahmad M. Virtual reality as a distraction technique for pain and anxiety among patients with breast cancer: A randomized control trial. Palliat Support Care. 2019 Feb;17(1):29-34. doi: 10.1017/S1478951518000639. Epub 2018 Sep 10. PMID 30198451
- [Background] Stevenson MP, Schilhab T, Bentsen P. Attention Restoration Theory II: a systematic review to clarify attention processes affected by exposure to natural environments. J Toxicol Environ Health B Crit Rev. 2018;21(4):227-268. doi: 10.1080/10937404.2018.1505571. Epub 2018 Aug 21. PMID 30130463
- [Background] Hartig T, Mang M, Evans GW. Restorative effects of natural environment experiences. Environ Behav. 1991;23:3-26.
- [Background] Li Y, Xing X, Shi X, Yan P, Chen Y, Li M, Zhang W, Li X, Yang K. The effectiveness of music therapy for patients with cancer: A systematic review and meta-analysis. J Adv Nurs. 2020 May;76(5):1111-1123. doi: 10.1111/jan.14313. Epub 2020 Feb 19. PMID 32017183
- [Background] Krishnaswamy P, Nair S. Effect of Music Therapy on Pain and Anxiety Levels of Cancer Patients: A Pilot Study. Indian J Palliat Care. 2016 Jul-Sep;22(3):307-11. doi: 10.4103/0973-1075.185042. PMID 27559260
- [Background] Lewis CH, Griffin MJ. Human factors consideration in clinical applications of virtual reality. Stud Health Technol Inform. 1997;44:35-56. PMID 10175342
- See also: NCCN Distress Thermometer and Problem List for Patients — https://www.nccn.org/docs/default-source/patient-resources/nccn_distress_thermometer.pdf?sfvrsn=ef1df1a2_4
- See also: Oculus Go warnings — https://www.meta.com/legal/quest/health-and-safety-warnings/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05690230/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT05690230/ICF_001.pdf